CLINICAL TRIAL: NCT01730521
Title: The Effect of a Short Term Exercise Schedule on Oral Iron Bio-availability and Iron Incorporation
Status: Completed | Type: Observational
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Professor, MD, Swiss Federal Institute of Technology
Other Study IDs: EK 2012-N-27
Record Dates: First submitted 2012-11-07; First posted 2012-11-21 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Generally Healthy
MeSH Terms: interventions — Exercise; Running

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Difference in Iron bioavailabilty exercise and resting phase: the subjects will act as their own control during the study
  Interventions: Behavioral: Exercise (Running)

INTERVENTIONS:
Behavioral: Exercise (Running) — the study foresees a measurement of iron biavailability in a resting and in a exercising phase and subjects will act as their own control during the study.

SUMMARY:
Iron metabolism may undergo changes during exercise, with reductions in classical iron status markers due to a variety of postulated mechanism which include hemodilution, increased iron loss, hemolysis and increased iron storage in muscles. Furthermore, it has been reported that vigorous training increases hepcidin, a central regulatory peptide in iron metabolism. This increase has been ascribed to the presence of subclinical inflammation. Increased hepcidin levels may reduce iron bioavailability and iron incorporation in erythrocytes.

Twenty healthy men subjects will be recruited as subjects for this study. Subjects should be generally healthy, with no history of blood donation in the last 6 months, should weigh less than 85 Kg, and not take iron supplements and/or multivitamin supplements. Subjects should have familiarity to sports and running, but not currently (i.e. in the past 3 months) training for more than 1h per week on average.

The aim of this study is to measure an iron bioavailability during a resting and an exercise phase lasting approx. 14 days with training sessions on alternate days. Subjects will participate in both restign and exercising protocols and act as their own controls during the study. Iron bioavailability will be measured via the incorporation of stable isotopic labels 14 days after administration. To control for changes in blood volume during the course of the study, blood volume of the participating subjects will be measured before and after the exercise phase with the CO-rebreathing method.

Measurement of iron bioavailability and iron incorporation in a resting and exercising phase will allow determine if the increased level of hepcidin seen in in exercise will induce a lower iron bioavailability and iron incorporation during exercise.

ELIGIBILITY:
Inclusion Criteria:

* men, Generally Healthy age between 18-50 years;
* BMI between 18-25;
* nonanemic (Hb < 120 g/L);
* no intake of vitamins and nutritional supplements;
* no recent blood donation (<4 months);
* no previous participation in studies with stable iron isotopes in the past.

Exclusion Criteria:

* Chronic diseases, Metabolic diseases, GI tract diseases (self reported)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects studying or working at the University of Zürich or ETH Zürich
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Iron bioavailability from Stable isotopic labels | Up to 2 months

SECONDARY OUTCOMES:
Blood volume increase during exercise | Up to 2 months

OTHER OUTCOMES:
Hepcidin levels and inflammation markers (C-Reactive Protein, 1-Alpha acid glycoprotein) | Up to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Diego Moretti, PhD, Principal Investigator — ETH Zürich
Locations (1):
- ETH Zürich, Zurich, Switzerland

REFERENCES:
- [Background] Cercamondi CI, Egli IM, Ahouandjinou E, Dossa R, Zeder C, Salami L, Tjalsma H, Wiegerinck E, Tanno T, Hurrell RF, Hounhouigan J, Zimmermann MB. Afebrile Plasmodium falciparum parasitemia decreases absorption of fortification iron but does not affect systemic iron utilization: a double stable-isotope study in young Beninese women. Am J Clin Nutr. 2010 Dec;92(6):1385-92. doi: 10.3945/ajcn.2010.30051. Epub 2010 Oct 6. PMID 20926522
- [Derived] Moretti D, Mettler S, Zeder C, Lundby C, Geurts-Moetspot A, Monnard A, Swinkels DW, Brittenham GM, Zimmermann MB. An intensified training schedule in recreational male runners is associated with increases in erythropoiesis and inflammation and a net reduction in plasma hepcidin. Am J Clin Nutr. 2018 Dec 1;108(6):1324-1333. doi: 10.1093/ajcn/nqy247. PMID 30351387